CLINICAL TRIAL: NCT02607020
Title: Self-Management Program Based on Physical Exercises for People With Multiple Sclerosis With Mild Neurological Impairment: A Randomized Controlled Trial
Brief Title: Self-Management Program Based on Physical Exercises in People With Multiple Sclerosis
Acronym: AUTOMOVEMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Hôpital Raymond Poincaré (Other); CHU de Reims (Other)
Responsible Party: Principal Investigator, Lejeune, professeur, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUTOMOVEMS01
Record Dates: First submitted 2015-11-09; First posted 2015-11-17 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Physical exercise (Experimental)
  Interventions: Other: Physical exercises in an self-management setting
- Relaxation (Active Comparator)
  Interventions: Other: Relaxation

INTERVENTIONS:
Other: Physical exercises in an self-management setting — Workout sessions will be based on the principle of self-management, without direct supervision of a therapist. Sessions will include:
  1. Twenty minutes of aerobic exercises 1.2. Five to ten minutes of stretching exercises. 2.3. Fifteen to twenty minutes of resistance exercises to improve muscle strength of lower limbs. The targeted muscles will be the hip flexors, the knee extensors and flexors, and the foot extensors and plantar flexors. These exercises will comply with the recommendations of the American College of Sports Medicine (ACSM, 2011). Patients will be asked to perform muscle contractions against the gravity (about 15 repeats). There will be on average 5 to 6 series per session. Several muscle groups of the lower limbs will be trained during the same session.
  Arms: Physical exercise
Other: Relaxation — The relaxation sessions of the control group will be carried out with the help of soothing music. Patients will receive a Compact Disc (CD) of soothing music at the inclusion. Patients will also have an electronic training logbook that will be reviewed each week by a therapist. They will have a phone contact with the therapist every two weeks, to discuss about the treatment and adapt it if necessary. They will also have a reminder session every four weeks.
  Arms: Relaxation

SUMMARY:
Fatigue is the most chronic and disabling symptom in multiple sclerosis patients. Self-management physical exercise programs seem promising to allow patients to improve their fatigue and their deconditioning. However, the effectiveness of such programs has been poorly assessed until now. The objectives of the present study are to evaluate the relationships between fatigue and physical capacity among slightly affected MS patients, and to carry on a large trial to assess the effectiveness of a self-management exercise program in the same patients. Sixty-four patients will be included and will be asked, after an educational period, to perform at least three exercise sessions of more than 30 minutes each week, over a period of three months. Patients will be splitted in two groups : one group will perform endurance and resistance physical exercises, and the other one will perform relaxation exercises with the help of soothing music. A regular coaching will adapt the exercises and motivate the patients to continue the treatment. Assessors won't be informed of patients' treatment. Four evaluations will be done, and will notably assess muscle strength, endurance, fatigue and social participation.

DETAILED DESCRIPTION:
Objectives: the aims of this project are two-fold:

* The first aim is to evaluate the relationships between fatigue and physical capacity, among multiple sclerosis (MS) patients at the early stage of the disease and their relations to plasmatic cytokines levels;
* The second aim is to assess the effectiveness of a self-management program of physiotherapy, based on endurance and resistance physical exercises, in MS patients at the early stage of the disease.

Rationale and scientific background:

Multiple sclerosis affects one person per thousand people in France and Belgium. Two thousand patients are newly diagnosed in France each year. Fatigue is an early and very disabling symptom of MS, that affects 50 to 80% of MS patients. Fatigue is described by patients as the most chronic and the most disabling symptom and is associated with a decline in motivation and a need for rest. Fatigue can occur spontaneously or can be induced by physical or mental activity, acute infection, or ingestion of food. It can occur at any time but usually worsens along the day.

Fatigue can have multiple origins in patients with MS: brain lesion load, cortical atrophy, dysfunction of the hypothalamo-pituitary axis, depression or physical deconditioning. Several approaches seem promising to improve fatigue: energy conservation programs, which help patients in organizing their daily activities to avoid fatigue, cognitive behavioural therapy, medications and physical exercise. Patients with MS show indeed a degradation of their cardio-respiratory endurance. This degradation seems to occur early in the course of MS, and to be already present in patients with mild neurological impairments. A deconditioning is regularly found in patients complaining of fatigue. However, the literature does not provide clear information about the relationship between physical deconditioning and fatigue, at the very early stage of MS.

Exercise medicine is therefore a promising approach in the management of fatigue. Several studies have shown an improvement of fatigue and gait ability after a program of physical exercise. Dalgas (2008) and Sandoval (2013) have proposed recommendations on endurance and resistance exercise in MS patients. Following their recommendations, endurance training should be made through walking or cycling exercise, 2 to 3 times per week, at an intensity corresponding to 60-80% of the predicted maximal heart rate. The recommended duration of sessions is 10 to 40 minutes, depending on patients' motor impairments. Resistance training should be preferentially supervised by therapists, at least for the first sessions. If the training is self-managed or home-based, using the weight of the body or elastic bands seems sufficient to bring an improvement in muscle strength. Three to four sets of exercises, separated by 2-4 minutes rest periods, with an intensity of 8 to 15 repetitions at 70% of the predicted maximum strength (RM), seem to be effective when carried out 2-3 times per week. Each program should include 4 to 8 various exercises. Few studies have rated the benefits of these programs in the long term and at the early stage of the disease. A precocious exercise prescription could prevent deconditioning or its effects, including fatigue.

Currently, a small number of patients benefits from physiotherapy treatments based on physical exercise. On one hand, multidisciplinary rehabilitation programs (including physiotherapy, occupational therapy, neuropsychology, physical exercise,...) are implemented only when impairments are severe (e.g. immediately after a relapse), due to the strict criteria of reimbursement established by social insurances. Therefore, patients who are only slightly impaired cannot benefit from these programs. Moreover, the lack of rehabilitation facilities allows only a limited number of patients to participate in multidisciplinary programs. On the other hand, few rehabilitation centres organize face-to-face or group-based physiotherapy programs specifically targeting physical exercise in patients with MS. Indeed, these face-to-face programs remain mainly focused on neurodevelopmental theories (Bobath,…). Finally, both multidisciplinary programs and specific exercise-based programs are mostly implemented in hospitals and large centres of rehabilitation. However, such structures do not seem necessary when the main objective is to do physical exercise, and can even be stressful for those patients with mild impairments.

An alternative to these treatments may be self-management physical exercise programs, supervised by physical medicine and rehabilitation teams. These programs only require a limited cost for the patient and the society, and can be done in an ecological environment (i.e. where the patient lives). These community-based rehabilitation programs could therefore enable a better adhesion to treatment than hospital treatments. The effectiveness of self-managed rehabilitation has poorly been assessed. Results of the literature are conflicting, and the evidence is lacking. These authors pointed the need for further randomised controlled trials.

The aim of our project is therefore to implement a physical exercise program in patients at the early stage of MS, including resistance and cardio-respiratory endurance exercises. A multicenter, single-blind, randomised controlled trial will be carried out to assess its effectiveness. This project will also study the fitness and fatigue in patients whose walking capacity is preserved.

It has also been noted that fatigue is related to the plasma levels of various cytokines (e.g. Interleukin(IL)-6, IL-10, Interferon-gamma(IFNg), Tumor Necrosis Factor-alpha (TNFa)...) and it has been suggested that physical exercise could reduce fatigue through an effect on the transcription of the genes coding for these cytokines.

In the following sections, the term "self-management program" will refer to the whole program, including education, exercises, and coaching of patients.

Research project:

This is a multicentre, single-blind, randomised controlled trial. All patients will initially have a consultation with an investigator for the screening visit, two weeks before inclusion. Inclusion and exclusion criteria will be checked, and a motivational interview of the patient will be done. Randomisation will also be carried out during this visit, and will be stratified to enable the equivalence of the Expanded Disability Status Scale (EDSS) scores in both the experimental and the control groups. The randomization will be separate for each center. The first evaluation will be performed the day of study inclusion (see below), by another investigator. A same investigator will carry out all assessment of a same patient. The second evaluation will take place two weeks later. Treatment will begin in the week following this evaluation for patients of both groups. No detailed information will be given to patients about the other group's treatment. They will only be informed that the aim of the study is to compare two rehabilitation treatments, one based on physical exercises and the other one based on relaxation.

Patients in the experimental group will participate in four two preliminary group-based educational sessions of one hour. The first session, a group-based session, will aim to explain the theoretical bases of physical exercise in MS disease (one hour). The next three session, a face-to-face interviews will be devoted to the demonstration and initial practice of the exercises that patients will have to perform during the self-management program (three one hours).

Patients will have an individual appointment of thirty minutes immediately after the last session, in order to define a program tailored to their individual goals. They will be asked to do at least three physical exercise sessions per week, more than forty-five minutes each, over a period of three months. The type of exercises and their intensity will be also specified to the patient on this occasion. These exercises will be carried out through a self-management program, and will then not be directly supervised by a therapist.

Patients in the control group will receive two four sessions (the first one in group and the second explaining how to practice relaxation with the help of soothing music (four two hours). They will then be invited to practice relaxation at home, for at least forty-five minutes per day, at least three times a week, over a period of three months.

Two Three last evaluations will be conducted in patients: one within the week after the end of the study, one six months after inclusion and one nine months after inclusion, in order to assess the long-term effects of the treatment.

At the end of the study (nine months after the inclusion), all patients of the control group will have the opportunity to benefit from a self-management program of exercises under indirect supervision, comparable to the treatment received by the experimental group during the study.

All patients will continue in parallel all other usual medical and paramedical treatments, including physiotherapy, these treatments remaining unchanged during this project.

Protocol of exercises:

see below

Patients will have access to a virtual training book on the internet, in which they will be asked to list all details about workouts within the hospital and at home (number, date, duration, exercises conducted, intensity). If some patients do not have access to the internet at home, a training logbook will be given at the inclusion, allowing them to list the exercises details at each session.

The training will be monitored each week through the electronic training book, by a therapist (physician or physical therapist), and recommendations on the self-management training will be conveyed by this virtual logbook. A phone contact between the patient and the therapist will be scheduled every two weeks. The patient will be encouraged to continue these exercises on a regular basis. Recommendations will be tailored to patient's capacity and to the exercises he will have been able to achieve the previous week. Every four weeks, a group-based reminder session will take place in the referring hospital, one for the experimental group and one for the control group, in order to check if there are some adverse effects, if exercises are performed correctly, and if the patient remains motivated for the continuation of support. The internet logbook of each patient will be reviewed on this occasion by the therapist in order to adapt exercises to the patient's capabilities and to the exercises carried out the previous weeks.

For patients who would have no internet at home, exercises will be followed and adapted each week from a telephone contact between the patient and a therapist, and from a consultation organised each two weeks to allow the therapist to examine the training book and to adapt the exercises if necessary.

The relaxation sessions of the control group will be carried out with the help of soothing music. Patients will receive a Compact Disc of soothing music at the inclusion. Patients will also have an electronic training logbook that will be reviewed each week by a therapist. They will have a phone contact with the therapist every two weeks, to discuss about the treatment and adapt it if necessary. They will also have a reminder session every four weeks.

Statistics:

Pearson and Spearman correlation coefficients will permit to study the relationships between fatigue and physical capacity. The calculation of the intraclass correlation coefficient will test the reproducibility of the two first evaluations. A two-factors analysis of variance (ANOVA) will be carried out to investigate the effectiveness of the self-management programs (Group X time). The Holm-Sidak test will be used as a post-hoc test.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of MS performed by a specialized neurologist (revised McDonald criteria, 2010), regardless of the form of the disease (relapsing-remitting, primary progressive, secondary progressive);
* An EDSS score less than or equal to 3.5, with a functional score less than or equal to 2 for the pyramidal and cerebellar functions;
* An age between 18 and 65 years.

Exclusion Criteria:

* An affection of one or both lower limbs limiting their ability to walk;
* Another illness contraindicating the practice of exercises (ACSM criteria, 2011);
* An episode of relapse within the 4 weeks prior to inclusion;
* Participation in a study targeting rehabilitation, within the 3 months prior to inclusion;
* Modification of drug treatment of MS (disease-modifying treatment and symptomatic treatment) in the 3 months prior to inclusion;
* Change in the physiotherapy prescription within the 3 months prior to inclusion.
* Pregnancy
* Participation in a regular exercise program at least 3 times a week for at least 30 minutes for more than 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 28 days
  Modified Fatigue Impact Scale (MFIS)
Change in fatigue | Evaluation at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  MFIS

SECONDARY OUTCOMES:
Safety (Number of patients with adverse events related to treatment). | Through study completion, an average of 9 months
  Number of patients with adverse events related to treatment
Change in MS-specific health related quality of life | 2 evaluations at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  Multiple Sclerosis Impact Scale (MSIS-29)
Change in MS-specific health related quality of life | 2 evaluations at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  Multiple Sclerosis International Quality of Life (MusiQol)
Change in walking capacity | 2 evaluations at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  using a questionnaire (MSWS-12)
Change in plasmatic cytokines: IFNg | Baseline and immediately after the intervention
  plasmatic titration of IFNg (pg/mL)
Change in plasmatic cytokines: TNFa | Baseline and immediately after the intervention
  plasmatic titration of TNFa (pg/mL)
Adherence | Weekly through the intervention (during 3 months)
  Percentage of sessions completed
Adherence | Weekly through the intervention (during 3 months)
  duration of exercising
Amount of physical activity performed | From the first day after the completion of the treatment, every 3 months up to 6 months.
  Using a self-reported questionnaire
Change in Cardiorespiratory fitness | 2 evaluations at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  physical working capacity at 75% of the predicted maximal heart rate per kilogram of body weight (PWC75%)
Change in Cardiorespiratory fitness | 2 evaluations at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  Oxygen Uptake Efficiency Slope (OUES)
Change in Lower limbs spasticity | 2 evaluations at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  Ashworth scale
Change in objective walking endurance | 2 evaluations at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  2 Minute Walking Test
Change in static and dynamic balance | 2 evaluations at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  Timed up-and-go test
Change in Neurological Disability | 2 evaluations at baseline, one immediately after the intervention program, one 3 months afterward and the last one 6 months after the end of the intervention
  Expanded Disability Status Scale

CONTACTS AND LOCATIONS:
Overall Officials: Maxime VALET, MD, Principal Investigator — UCL
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Background] Baert I, Freeman J, Smedal T, Dalgas U, Romberg A, Kalron A, Conyers H, Elorriaga I, Gebara B, Gumse J, Heric A, Jensen E, Jones K, Knuts K, Maertens de Noordhout B, Martic A, Normann B, Eijnde BO, Rasova K, Santoyo Medina C, Truyens V, Wens I, Feys P. Responsiveness and clinically meaningful improvement, according to disability level, of five walking measures after rehabilitation in multiple sclerosis: a European multicenter study. Neurorehabil Neural Repair. 2014 Sep;28(7):621-31. doi: 10.1177/1545968314521010. Epub 2014 Feb 6. PMID 24503204
- [Background] Batcho CS, Thonnard JL, Nielens H. PWC 75%/kg, a fitness index not linked to resting heart rate: testing procedure and reference values. Arch Phys Med Rehabil. 2012 Jul;93(7):1196-200. doi: 10.1016/j.apmr.2012.02.021. Epub 2012 Mar 8. PMID 22521927
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Boudarham J, Roche N, Pradon D, Delouf E, Bensmail D, Zory R. Effects of quadriceps muscle fatigue on stiff-knee gait in patients with hemiparesis. PLoS One. 2014 Apr 9;9(4):e94138. doi: 10.1371/journal.pone.0094138. eCollection 2014. PMID 24718087
- [Background] Cakt BD, Nacir B, Genc H, Saracoglu M, Karagoz A, Erdem HR, Ergun U. Cycling progressive resistance training for people with multiple sclerosis: a randomized controlled study. Am J Phys Med Rehabil. 2010 Jun;89(6):446-57. doi: 10.1097/PHM.0b013e3181d3e71f. PMID 20216060
- [Background] Carter A, Daley A, Humphreys L, Snowdon N, Woodroofe N, Petty J, Roalfe A, Tosh J, Sharrack B, Saxton JM. Pragmatic intervention for increasing self-directed exercise behaviour and improving important health outcomes in people with multiple sclerosis: a randomised controlled trial. Mult Scler. 2014 Jul;20(8):1112-22. doi: 10.1177/1352458513519354. Epub 2014 Jan 13. PMID 24421303
- [Background] Cattaneo D, Regola A, Meotti M. Validity of six balance disorders scales in persons with multiple sclerosis. Disabil Rehabil. 2006 Jun 30;28(12):789-95. doi: 10.1080/09638280500404289. PMID 16754576
- [Background] Dalgas U, Stenager E, Ingemann-Hansen T. Multiple sclerosis and physical exercise: recommendations for the application of resistance-, endurance- and combined training. Mult Scler. 2008 Jan;14(1):35-53. doi: 10.1177/1352458507079445. Epub 2007 Sep 19. PMID 17881393
- [Background] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Resistance training improves muscle strength and functional capacity in multiple sclerosis. Neurology. 2009 Nov 3;73(18):1478-84. doi: 10.1212/WNL.0b013e3181bf98b4. PMID 19884575
- [Background] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458
- [Background] Giovannoni G. Multiple sclerosis related fatigue. J Neurol Neurosurg Psychiatry. 2006 Jan;77(1):2-3. doi: 10.1136/jnnp.2005.074948. PMID 16361582
- [Background] Goldman MD, Marrie RA, Cohen JA. Evaluation of the six-minute walk in multiple sclerosis subjects and healthy controls. Mult Scler. 2008 Apr;14(3):383-90. doi: 10.1177/1352458507082607. Epub 2007 Oct 17. PMID 17942508
- [Background] Guerra E, di Cagno A, Mancini P, Sperandii F, Quaranta F, Ciminelli E, Fagnani F, Giombini A, Pigozzi F. Physical fitness assessment in multiple sclerosis patients: a controlled study. Res Dev Disabil. 2014 Oct;35(10):2527-33. doi: 10.1016/j.ridd.2014.06.013. Epub 2014 Jul 5. PMID 25000308
- [Background] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714
- [Background] Induruwa I, Constantinescu CS, Gran B. Fatigue in multiple sclerosis - a brief review. J Neurol Sci. 2012 Dec 15;323(1-2):9-15. doi: 10.1016/j.jns.2012.08.007. Epub 2012 Aug 27. PMID 22935407
- [Background] Krupp L. Fatigue is intrinsic to multiple sclerosis (MS) and is the most commonly reported symptom of the disease. Mult Scler. 2006 Aug;12(4):367-8. doi: 10.1191/135248506ms1373ed. No abstract available. PMID 16900749
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Background] Lauer RT, Stackhouse C, Shewokis PA, Smith BT, Orlin M, McCarthy JJ. Assessment of wavelet analysis of gait in children with typical development and cerebral palsy. J Biomech. 2005 Jun;38(6):1351-7. doi: 10.1016/j.jbiomech.2004.07.002. PMID 15863120
- [Background] Nilsagard Y, Lundholm C, Gunnarsson LG, Dcnison E. Clinical relevance using timed walk tests and 'timed up and go' testing in persons with multiple sclerosis. Physiother Res Int. 2007 Jun;12(2):105-14. doi: 10.1002/pri.358. PMID 17536648
- [Background] Heine M, van de Port I, Rietberg MB, van Wegen EE, Kwakkel G. Exercise therapy for fatigue in multiple sclerosis. Cochrane Database Syst Rev. 2015 Sep 11;2015(9):CD009956. doi: 10.1002/14651858.CD009956.pub2. PMID 26358158
- [Background] Plow MA, Finlayson M, Rezac M. A scoping review of self-management interventions for adults with multiple sclerosis. PM R. 2011 Mar;3(3):251-62. doi: 10.1016/j.pmrj.2010.11.011. PMID 21402370
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Rae-Grant AD, Turner AP, Sloan A, Miller D, Hunziker J, Haselkorn JK. Self-management in neurological disorders: systematic review of the literature and potential interventions in multiple sclerosis care. J Rehabil Res Dev. 2011;48(9):1087-100. doi: 10.1682/jrrd.2010.08.0159. PMID 22234713
- [Background] Rossier P, Wade DT. Validity and reliability comparison of 4 mobility measures in patients presenting with neurologic impairment. Arch Phys Med Rehabil. 2001 Jan;82(1):9-13. doi: 10.1053/apmr.2001.9396. PMID 11239279
- [Background] Sandoval AE. Exercise in multiple sclerosis. Phys Med Rehabil Clin N Am. 2013 Nov;24(4):605-18. doi: 10.1016/j.pmr.2013.06.010. Epub 2013 Aug 2. PMID 24314679
- [Background] Simeoni M, Auquier P, Fernandez O, Flachenecker P, Stecchi S, Constantinescu C, Idiman E, Boyko A, Beiske A, Vollmer T, Triantafyllou N, O'Connor P, Barak Y, Biermann L, Cristiano E, Atweh S, Patrick D, Robitail S, Ammoury N, Beresniak A, Pelletier J; MusiQol study group. Validation of the Multiple Sclerosis International Quality of Life questionnaire. Mult Scler. 2008 Mar;14(2):219-30. doi: 10.1177/1352458507080733. Epub 2007 Oct 17. PMID 17942521
- [Background] Vernay D, Gerbaud L, Biolay S, Coste J, Debourse J, Aufauvre D, Beneton C, Colamarino R, Glanddier PY, Dordain G, Clavelou P. [Quality of life and multiple sclerosis: validation of the french version of the self-questionnaire (SEP-59)]. Rev Neurol (Paris). 2000 Mar;156(3):247-63. French. PMID 10740096
- [Background] Wade DT. Measurement in neurological rehabilitation. Curr Opin Neurol Neurosurg. 1992 Oct;5(5):682-6. PMID 1392142
- [Background] Yusuf A, Koski L. A qualitative review of the neurophysiological underpinnings of fatigue in multiple sclerosis. J Neurol Sci. 2013 Jul 15;330(1-2):4-9. doi: 10.1016/j.jns.2013.04.012. Epub 2013 May 4. PMID 23651867
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820